CLINICAL TRIAL: NCT00590434
Title: The Yield and Safety of Screening and Surveillance Colonoscopy in Elderly Patients (> 80 Years)
Brief Title: Yield and Safety of Colonoscopy in Patients Older Than 80 Years
Status: Completed | Type: Observational
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ajay Bansal, Principal Investigator, Staff Physician, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Other Study IDs: AB0002
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Neoplasms
Keywords: CRC - Colorectal cancer; CVA - Cerebral Vascular Accident; MI - Myocardial Infarction; CAD - Coronary Artery Disease; DM - Diabetes Mellitus; PVD - Peripheral Vascular Disease; NSAIDS - Non-Steroidal Anti inflammatory Drugs; screening; colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Stroke; Myocardial Infarction; Coronary Artery Disease; Diabetes Mellitus; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients older than 80 years presenting for average risk screening or surveillance colonoscopy
- 2: Patients younger than 80 years presenting for average risk screening or surveillance colonoscopy

SUMMARY:
The aim of the study is to study the risk of colorectal cancer and polyps in people older than 80 years compared to the younger age group. The researchers hypothesized that colonoscopy in older people is likely to have more complications without detection of a significant number of large polyps and cancer.

DETAILED DESCRIPTION:
Background and Clinical Significance:

Colorectal cancer continues to carry a significant burden of morbidity and mortality into the twenty-first century, despite the availability of multiple screening modalities. It is estimated that approximately 150,000 new cases of CRC will be diagnosed and over 50,000 people will die of CRC in 2006 (1). Current options for screening for CRC include fecal occult-blood testing, flexible sigmoidoscopy, double contrast barium enema, and colonoscopy. While no randomized controlled trials have shown a mortality benefit with screening colonoscopy, it has become the preferred method of both screening and surveillance of polyps because of the ability to visualize the entire colon in addition to having the ability to remove polyps. This procedure does associated risks including perforation and bleeding after polypectomy. Other major complications have also been reported, including MI and CVA.

Although guidelines exist for colorectal cancer screening and surveillance of polyps, they do not define the upper age limit to which these practices should be carried out (2,3). No clear data is available on the effect of this procedure on life expectancy after the age of 80. Also, the country has limited resources and screening colonoscopy may be offered to those who are most likely to benefit. Based on these facts, there is a real need to quantify the prevalence of colon neoplasia in this age group to guide primary care physicians as well as gastroenterologists in offering screening and surveillance colonoscopy to this age group. Like many medical decisions, cancer screening requires weighing quantitative information, such as risk of cancer death and likelihood of beneficial and adverse screening outcomes, as well as qualitative factors, such as individual patients' values and preferences. In fact, patients with life expectancies of less than 5 years are unlikely to derive any survival benefit from cancer screening. There is also potential for harm from screening procedures. Some of the greatest harms of screening occur by detecting cancers that would never have become clinically significant. This becomes more likely as life expectancy decreases.

As the population ages and life expectancy continues to increase, more elderly patients will be referred for colonoscopy. What is the utility of performing colonoscopy in these asymptomatic patients, and is it safe? Few studies have examined this question adequately. What follows is a brief review of published data in regards to yield and safety of colonoscopy in the elderly.

Yield:

Lin et al examined the prevalence of neoplasia in 1244 screening colonoscopies - 63 were patients older than 80. They found that although the prevalence of neoplasia increases with age (28.6% in patients older than 80), the gain in expected life expectancy after intervention is limited (4).

Cooper et al came to a somewhat different conclusion (7). They analyzed 1.8 million Medicare patient colonoscopies in 1999 using ICD-9 codes for rates of polyp detection (pathology was not examined, so it is not clear what percentage of these patients had hyperplastic polyps, adenomas, advanced adenomas, or cancer). They found that the rate of polyp detection decreased with age but was still high (ranging from 15.2-31.3% in patients older than 80). Cooper had previously shown that the incidence of colorectal cancer increased with age in an analysis of all new cases of colon cancer in Medicare patients in 19878. Similarly, the National Polyp Study has shown an increase in the incidence of high grade dysplasia in patients older than 60 (9).

Finally, the VA Cooperative Study Group No. 380 did a prospective cross sectional study of 3121 asymptomatic patients between 1994-1997 to find the prevalence of advanced neoplasia and associated risk factors. 329 patients were found to have advanced neoplasia as defined by an adenoma greater than 1 cm, villous histology, presence of high-grade dysplasia, or cancer. Associations were found between advanced neoplasia and family history of CRC, smoking, moderate to heavy alcohol consumption, fiber intake, and use of daily NSAIDS or vitamin D11.

Safety:

Two of the above studies discussed safety of colonoscopy in elderly patients. Duncan found 8 major complications (0.6%) including 3 bleeds and 1 perforation in a series of 1199 colonoscopies6. Sardinha also reported a low rate of major bleeding (0.2%) and no perforation in 428 colonoscopies; this compared favorably with two other studies on elderly patients.10 Gatto et al took a random sample of Medicare patients who underwent a colonoscopy between 1991 and 1998. 39,286 colonoscopies were identified by CPT-4 codes; perforations within 7 days of the procedure were identified by ICD-9 codes. The average age was 74, and 21 % of patients were older than 80. The overall incidence of perforation was 0.19%; the authors found that the rate of perforation increased with age and the number of comorbidities12,13.

In addition to perforation and bleeding, MI and CVA have also been reported after colonoscopy. Cappell studied patients who were already at higher risk for an MI or CVA. He looked at 100 patients who underwent colonoscopy within 30 days after MI and compared them to 100 control patients without MI or unstable angina in the preceding 6 months. He found that while there was a higher rate of minor complications (transient asymptomatic hypotension or bradycardia) in the study group (in which the patients were sicker overall), there was only one major complication after colonoscopy which was probably not due to the procedure13.

Importance of Current Research to Veterans:

The prevalence of CRC is approximately 5% (1,3). Although over 80% of cases are sporadic (the remaining result from inflammatory bowel disease and hereditary colon cancer syndromes), many veterans have one or more risk factors for CRC including advancing age, smoking, heavy alcohol intake, high fat low fiber diet, sedentary lifestyle, and obesity. As the veteran population ages, preventative services will continue to be an important part of their health care. As the US population is aging, so too is the US veteran population. This is further complicated by the fact that a recent study that examined the self-rated health and functioning of a national sample of veterans aged 65 or older reported that over one-half of elderly veterans report difficulty in functioning and rated their health status as fair or poor (14). This group of veterans may also live alone, may not have easy access to transportation to and from a health facility and may find it physically challenging to prepare their colon with cleansing agents for a good exam during a colonoscopy. Age and comorbidity also affect the survival rates after resection of colorectal cancer. A study by Ko et al used nationwide data from the healthcare cost and utilization program and calculated mortality among 22,000 resections for colon cancer15. They found that besides the volume of surgery, two other factors that affect post colon cancer mortality are age and comorbid disease (i.e. cardiovascular, pulmonary and liver diseases) (p<0.05). Another study of 80 patients (16), 80 years and older, showed a postoperative mortality rate of 8% and 5yr survival of only 23%. Only 13 patients lived longer than 5 years. Many elderly people may need a coronary revascularization procedure before planned surgery, if a colon cancer is discovered. Older age has been associated with adverse outcomes in patients undergoing percutaneous coronary intervention. A study by the National Heart, Lung and Blood Institute included 4620 PCI treated patients and reported adjusted relative risks in elderly (>80 years) compared to younger (<65 years) patients to be higher for inhospital related death (3.64 versus 1.0) as well as myocardial infarction (2.57 versus 1.0) (17).

Based on the above data, it is useful and necessary to know the potential risks and benefits of this invasive procedure in otherwise asymptomatic elderly patients.

Methods:

Study Design: Computerized medical records and endoscopy reports will be searched to identify patients older than 80 years old who underwent colonoscopy indicated for average risk screening for colon cancer or surveillance of polyps. A control group of patients between the ages of 50 and 79 will also be identified who underwent colonoscopy indicated for average risk screening for colon cancer or surveillance of polyps. The ratio of controls to study patients will be 2 to 1. Records will be searched from 1997 to July 31, 2006. Data collected will include age at time of colonoscopy, sex, body mass index, a personal history of CAD, DM, CVA, or PVD, endoscopic and histologic findings of colonoscopy, evidence of complete examination, all complications during colonoscopy, evidence of complications after colonoscopy including perforation, bleeding, MI, and CVA. The use of aspirin, NSAIDS, calcium, and vitamin D will be recorded. A comprehensive questionnaire that will include information on diet, exercise, family history, smoking, alcohol consumption, use of aspirin, NSAIDS, calcium, vitamin D, and statins will be administered by the endoscopist prior to colonoscopy.

Risk and Benefit to the Study Participant:

The participants will only be active in the prospective portion of the study. Their participation will be limited to completion of a written survey. This will be given after verbal informed consent. There will be no risk to the study participant. Benefits of this study have been previously addressed in detail in the section titled " Importance of Current Research to Veterans".

Data Collection:

Patient demographics, endoscopy and pathology findings, procedure complications, comorbidities and data regarding various risk factors such as smoking, alcohol intake, lack of dietary fruits and vegetables, lack of exercise, family history, prior history of colon cancer, ASA, NSAID and statin use will be collected. A questionnaire for the factors outlined above will be administered by an endoscopist. The data will be transferred to an Excel spreadsheet by one of the study investigators.

Statistical Power and Data Analysis:

Using the SPSS software, the prevalence of colon polyps and colon cancer between the group age >80 years and < 80 years will be compared. Significant polyps will be defined as polyp > 1 cm in size, polyps with villous histology, three or more polyps and polyps with dysplasia. Hyperplastic polyps will be considered non-neoplastic. Smokers will be defined as people who smoked at least 1 pack per day for 10 years and who did not quit smoking in the past 10 years. Associations between the clinical and demographic variables will be examined using Spearman's correlation coefficients. Univariate analysis will be performed Chi-square or fisher's exact test for categorical variables and Wilcoxon sum test for continuous variables. A multivariate logistic regression will be performed to control for the covariates that may affect the prevalence of colonic neoplasia. All tests will be two-tailed. A p value of < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for colonoscopy after 1997
* Age 80 or older for the study group
* Age 50-79 for the control group
* Indications for colonoscopy:
* Average risk screening for CRC
* Surveillance of polyps (tubular adenomas)

Exclusion Criteria:

* Any colonoscopy done for symptoms (abdominal pain, weight loss, hematochezia, occult blood in stool, etc) or signs (iron deficiency anemia)
* Patients who are not average risk based on family history of CRC
* Diagnosis of ulcerative colitis or Crohn's Disease
* History of CRC
* Exams that were not completed to the cecum (except in cases of obstructing masses found to be neoplastic) or poor bowel preparation limiting visualization of the mucosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is a Veteran population presenting to a VA Hospital upper endoscopy unit
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2006-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Proportion of elderly patients (>80 yrs) with colorectal neoplasia | 2 years
proportion of patients with complications including perforation, bleeding, MI or CVA within 24 hours of colonoscopy in >80 vs. <80 agr group | 2 years

SECONDARY OUTCOMES:
Five year disease free survival and five year mortality rates after the diagnosis of colon cancer in older (>80 yrs) vs. younger group (<80 yrs) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Bansal, MD, Principal Investigator — Kansas City VA Medical Center
Locations (1):
- Kansascity VA Medical center, Kansas City, Missouri, United States

REFERENCES:
- [Background] Winawer S, Fletcher R, Rex D, Bond J, Burt R, Ferrucci J, Ganiats T, Levin T, Woolf S, Johnson D, Kirk L, Litin S, Simmang C; Gastrointestinal Consortium Panel. Colorectal cancer screening and surveillance: clinical guidelines and rationale-Update based on new evidence. Gastroenterology. 2003 Feb;124(2):544-60. doi: 10.1053/gast.2003.50044. PMID 12557158
- [Background] Winawer SJ, Zauber AG, Fletcher RH, Stillman JS, O'Brien MJ, Levin B, Smith RA, Lieberman DA, Burt RW, Levin TR, Bond JH, Brooks D, Byers T, Hyman N, Kirk L, Thorson A, Simmang C, Johnson D, Rex DK; US Multi-Society Task Force on Colorectal Cancer; American Cancer Society. Guidelines for colonoscopy surveillance after polypectomy: a consensus update by the US Multi-Society Task Force on Colorectal Cancer and the American Cancer Society. Gastroenterology. 2006 May;130(6):1872-85. doi: 10.1053/j.gastro.2006.03.012. PMID 16697750
- [Background] Lin OS, Kozarek RA, Schembre DB, Ayub K, Gluck M, Drennan F, Soon MS, Rabeneck L. Screening colonoscopy in very elderly patients: prevalence of neoplasia and estimated impact on life expectancy. JAMA. 2006 May 24;295(20):2357-65. doi: 10.1001/jama.295.20.2357. PMID 16720821
- [Background] Stevens T, Burke CA. Colonoscopy screening in the elderly: when to stop? Am J Gastroenterol. 2003 Aug;98(8):1881-5. doi: 10.1111/j.1572-0241.2003.07576.x. PMID 12907348
- [Background] Duncan JE, Sweeney WB, Trudel JL, Madoff RD, Mellgren AF. Colonoscopy in the elderly: low risk, low yield in asymptomatic patients. Dis Colon Rectum. 2006 May;49(5):646-51. doi: 10.1007/s10350-005-0306-3. PMID 16482421
- [Background] Cooper GS, Chak A, Koroukian S. The polyp detection rate of colonoscopy: a national study of Medicare beneficiaries. Am J Med. 2005 Dec;118(12):1413. doi: 10.1016/j.amjmed.2005.06.019. PMID 16378787
- [Background] Cooper GS, Yuan Z, Landefeld CS, Johanson JF, Rimm AA. A national population-based study of incidence of colorectal cancer and age. Implications for screening in older Americans. Cancer. 1995 Feb 1;75(3):775-81. doi: 10.1002/1097-0142(19950201)75:33.0.co;2-d. PMID 7828127
- [Background] O'Brien MJ, Winawer SJ, Zauber AG, Gottlieb LS, Sternberg SS, Diaz B, Dickersin GR, Ewing S, Geller S, Kasimian D, et al. The National Polyp Study. Patient and polyp characteristics associated with high-grade dysplasia in colorectal adenomas. Gastroenterology. 1990 Feb;98(2):371-9. PMID 2403953
- [Background] Sardinha TC, Nogueras JJ, Ehrenpreis ED, Zeitman D, Estevez V, Weiss EG, Wexner SD. Colonoscopy in octogenarians: a review of 428 cases. Int J Colorectal Dis. 1999 Aug;14(3):172-6. doi: 10.1007/s003840050205. PMID 10460909
- [Background] Lieberman DA, Prindiville S, Weiss DG, Willett W; VA Cooperative Study Group 380. Risk factors for advanced colonic neoplasia and hyperplastic polyps in asymptomatic individuals. JAMA. 2003 Dec 10;290(22):2959-67. doi: 10.1001/jama.290.22.2959. PMID 14665657
- [Background] Gatto NM, Frucht H, Sundararajan V, Jacobson JS, Grann VR, Neugut AI. Risk of perforation after colonoscopy and sigmoidoscopy: a population-based study. J Natl Cancer Inst. 2003 Feb 5;95(3):230-6. doi: 10.1093/jnci/95.3.230. PMID 12569145
- [Background] Cappell MS. Safety and efficacy of colonoscopy after myocardial infarction: an analysis of 100 study patients and 100 control patients at two tertiary cardiac referral hospitals. Gastrointest Endosc. 2004 Dec;60(6):901-9. doi: 10.1016/s0016-5107(04)02277-1. PMID 15605004
- [Background] Villa VM, Harada ND, Washington D, Damron-Rodriguez J. The health and functional status of US veterans aged 65+: implications for VA health programs serving an elderly, diverse veteran population. Am J Med Qual. 2003 May-Jun;18(3):108-16. doi: 10.1177/106286060301800304. PMID 12836900
- [Background] Ko CY, Chang JT, Chaudhry S, Kominski G. Are high-volume surgeons and hospitals the most important predictors of in-hospital outcome for colon cancer resection? Surgery. 2002 Aug;132(2):268-73. doi: 10.1067/msy.2002.125721. PMID 12219022
- [Background] Houry S, Amenabar J, Rezvani A, Huguier M. Should patients over 80 years old be operated on for colorectal or gastric cancer? Hepatogastroenterology. 1994 Dec;41(6):521-5. PMID 7536703
- [Background] Cohen HA, Williams DO, Holmes DR Jr, Selzer F, Kip KE, Johnston JM, Holubkov R, Kelsey SF, Detre KM; NHLBI Dynamic Registry. Impact of age on procedural and 1-year outcome in percutaneous transluminal coronary angioplasty: a report from the NHLBI Dynamic Registry. Am Heart J. 2003 Sep;146(3):513-9. doi: 10.1016/S0002-8703(03)00259-X. PMID 12947372
- [Background] Clipp EC, Carver EH, Pollak KI, Puleo E, Emmons KM, Onken J, Farraye FA, McBride CM. Age-related vulnerabilities of older adults with colon adenomas: evidence from Project Prevent. Cancer. 2004 Mar 1;100(5):1085-94. doi: 10.1002/cncr.20082. PMID 14983506
- [Background] Chen H, Cantor A, Meyer J, Beth Corcoran M, Grendys E, Cavanaugh D, Antonek S, Camarata A, Haley W, Balducci L, Extermann M. Can older cancer patients tolerate chemotherapy? A prospective pilot study. Cancer. 2003 Feb 15;97(4):1107-14. doi: 10.1002/cncr.11110. PMID 12569613
- [Background] Neagoe A, Molnar AM, Acalovschi M, Seicean A, Serban A. Risk factors for colorectal cancer: an epidemiologic descriptive study of a series of 333 patients. Rom J Gastroenterol. 2004 Sep;13(3):187-93. PMID 15470530
- [Background] Anderson JC, Alpern Z, Messina CR, Lane B, Hubbard P, Grimson R, Ells PF, Brand DL. Predictors of proximal neoplasia in patients without distal adenomatous pathology. Am J Gastroenterol. 2004 Mar;99(3):472-7. doi: 10.1111/j.1572-0241.2004.04093.x. PMID 15056088
- [Background] Juarranz M, Calle-Puron ME, Gonzalez-Navarro A, Regidor-Poyatos E, Soriano T, Martinez-Hernandez D, Rojas VD, Guinee VF. Physical exercise, use of Plantago ovata and aspirin, and reduced risk of colon cancer. Eur J Cancer Prev. 2002 Oct;11(5):465-72. doi: 10.1097/00008469-200210000-00009. PMID 12394244
- [Background] Terry MB, Neugut AI, Mansukhani M, Waye J, Harpaz N, Hibshoosh H. Tobacco, alcohol, and p53 overexpression in early colorectal neoplasia. BMC Cancer. 2003 Nov 6;3:29. doi: 10.1186/1471-2407-3-29. PMID 14604438
- [Background] Thun MJ, Namboodiri MM, Heath CW Jr. Aspirin use and reduced risk of fatal colon cancer. N Engl J Med. 1991 Dec 5;325(23):1593-6. doi: 10.1056/NEJM199112053252301. PMID 1669840
- [Background] Poynter JN, Gruber SB, Higgins PD, Almog R, Bonner JD, Rennert HS, Low M, Greenson JK, Rennert G. Statins and the risk of colorectal cancer. N Engl J Med. 2005 May 26;352(21):2184-92. doi: 10.1056/NEJMoa043792. PMID 15917383
- See also: NCI Colorectal statistics — http://www.seer.cancer.gov/statfacts/html/colorect.html